CLINICAL TRIAL: NCT05841745
Title: Multicenter Registry on Robotically Assisted Percutaneous Coronary Interventions - TESLA Registry
Brief Title: Multicenter Registry on Robotically Assisted PCI - TESLA
Acronym: TESLA
Status: Recruiting | Type: Observational
Sponsor: Clinical Research Center, Intercard Sp. z o.o. (Industry)
Collaborators: Corindus, Inc. dba Siemens Healthineers Endovascular Robotics (Unknown); KCRI Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Other Study IDs: TESLA Protocol Version 2.1
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Robotically-assisted percutaneous coronary intervention; Coronary artery disease; R-PCI registry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Robotically-Assisted Percutaneous Coronary Intervention: All patients older than 18 years, who underwent R-PCI (defined as completion of at least one procedural step robotically) with the CorPath GRX System (Corindus Vascular) and completed one-year follow-up including patients with either stable coronary artery disease, unstable angina, or acute myocardial infarction (MI).
  Interventions: Device: Robotically-Assisted Percutaneous Coronary Intervention with CorPath GRX System

INTERVENTIONS:
Device: Robotically-Assisted Percutaneous Coronary Intervention with CorPath GRX System — The CorPath GRX System is intended for use in the remote delivery and manipulation of guidewires and rapid exchange catheters, and remote manipulation of guide catheters during percutaneous coronary and vascular procedures. The CorPath GRX System is composed of two units; the first is a bedside unit which consists of the extended robotic arm, robotic drive, and single-use loading cassette, and the second is the remote workstation, which consists of the interventional cockpit and the control console. A key innovation of the CorPath GRX System is the software-based automation of common maneuvers, called technIQ automated movements with the potential to increase procedural success, reduce procedure time, and generally increase user comfort with robotic assistance during PCI.

SUMMARY:
MulTicenter rEgiStry on RoboticalLy Assisted percutaneous coronary interventions- TESLA registry is a retrospective registry evaluating the safety and efficacy of robotically assisted PCI with the CorPath GRX System (Corindus Vascular, Siemens Healthineers, Germany) in real-world interventional cardiology practice.

DETAILED DESCRIPTION:
R-PCI represents a novel approach to performing PCI with several studies showing high technical success and low complication rates. The CorPath GRX System is the second generation of the CorPath platform, dedicated to advancing robotic-assisted vascular procedures to mitigate the orthopaedic and radiation-related occupational hazards associated with the practice of interventional cardiology.

MulTicenter rEgiStry on RoboticalLy Assisted percutaneous coronary interventions- TESLA registry is a retrospective registry evaluating the safety and efficacy of robotically assisted PCI with the CorPath GRX System (Siemens Healthineers, Germany) in real-world interventional cardiology practice in Europe and Asia.

All patients who underwent R-PCI (defined as completion of at least one procedural step robotically) with the CorPath GRX System and completed one-year follow-up are eligible for recruitment in this registry, if older than 18 years. This study includes patients with either stable coronary artery disease, unstable angina, or acute myocardial infarction (MI).

The Study Investigators expect to enroll at least 700 patients (up to 1000). International centers that performed R-PCI with the CorPath GRX System will be invited to participate in this multicenter study.

Baseline, procedural, and follow-up data will be collected for all cases.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years,
* Patients with either stable coronary artery disease, unstable angina, or acute myocardial infarction (MI),
* Coronary artery lesions considered suitable for R-PCI with CorPath GRX System.

Exclusion Criteria:

- Unwillingness to provide informed consent (only if applicable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry will include at least 700 patients (up to 1000) who underwent R-PCI. All the international centers that have already utilized the CorPath GRX System have been invited to participate in this multicenter study. The final number of patients enrolled in the study will depend on the final number of participating centers and the number of patients treated with R-PCI with CorPath GRX System in each center. All patients who underwent R-PCI (defined as completion of at least one procedural step robotically) with the CorPath GRX System (Corindus Vascular) and completed one-year follow-up are eligible for recruitment in this registry, if older than 18 years. This study includes patients with either stable coronary artery disease, unstable angina, or acute myocardial infarction (MI).
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinically successful PCI | From time of procedure until date of first event or death from any cause, which came first, assessed up to the time of discharge in the index hospitalization
  Clinical success, defined as angiographic success (residual stenosis after stenting of <30% with final TIMI [Thrombolysis In Myocardial Infarction] flow grade 3) without an in-hospital major adverse cardiovascular event (MACE) (death, target vessel MI, or need of repeat target vessel revascularization);

SECONDARY OUTCOMES:
Number of participants with ischemia-driven target lesion revascularization (TLR) | 1 year post-procedure
  Ischemia-driven target lesion revascularization (TLR), at 1 year defined according to the Academic Research Consortium (ARC) criteria;
Number of participants with target lesion failure (TLF) | 1 year post-procedure
  Target lesion failure (TLF) at 1 year, the composite of ARC-defined cardiac death, target vessel MI, or ischemia-driven TLR;
Number of participants with target vessel failure (TVF) | 1 year post-procedure
  Target vessel failure (TVF) at 1 year, the composite of ARC-defined cardiac death, target vessel MI, or ischemia-driven TVR.
Procedure time | During the procedure
  The time recorded from initial guidewire insertion into the robotic drive until guide catheter disengagement.
Contrast volume | During the procedure
  The total contrast volume used during the procedure.
Patient radiation exposure | During the procedure
  Dose-area-product (DAP) as recorded during the procedure.

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE) | From time of procedure until date of first event or death from any cause, which came first, assessed up to the time of discharge in the index hospitalization
  In-hospital MACE, the composite of death, target vessel MI, or need of repeat target vessel revascularization;
Number of participants with stent thrombosis | 1 year post-procedure
  Stent thrombosis at 1 year, defined according to the ARC criteria;
Bleeding events | 1 year post-procedure
  Bleeding events at 1 year, defined according to the Bleeding ARC (BARC).
Manual input and/or conversion | During the procedure
  The incidence and reasons for manual input and/or conversion during R-PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, PhD, Principal Investigator — Clinical Research Center Intercard
Locations (6):
- Hartcentrum OLV Aalst, Aalst, Belgium
- Germany (2):
  - SEGEBERGER Kliniken GmbH, Bad Segeberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
- Sapporo Cardiovascular Clinic, Sapporo, Japan
- Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Nowy Sącz, Malopolska, Poland
- Hospital Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No